CLINICAL TRIAL: NCT06064539
Title: A Phase 1, Single-center, Open-label, Two-cohort, Two-period, One-sequence, Two Treatment, Drug-drug Interaction Study of the Effects of Gemfibrozil and Rifampicin on SAR442168 in Healthy Subjects
Brief Title: Study of Drug-drug Interaction of the Effects of Gemfibrozil and Rifampicin on SAR442168 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INT16726; U1111-1244-2759 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Gemfibrozil; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): SAR442168 administered alone and together with gemfibrozil. 1 day washout for each administration of SAR442168.
  Interventions: Drug: Tolebrutinib; Drug: gemfibrozil
- Cohort 2 (Experimental): SAR442168 administered alone and together with rifampicin. 1 day washout for each administration of SAR442168.
  Interventions: Drug: Tolebrutinib; Drug: rifampicin

INTERVENTIONS:
Drug: Tolebrutinib — Tablet, taken orally
Drug: gemfibrozil — Tablet, taken orally
  Arms: Cohort 1
Drug: rifampicin — Tablet, taken orally
  Arms: Cohort 2

SUMMARY:
This is a Phase 1, single-center, open-label, non-randomized study to assess the effects of CYP2C8 inhibition using gemfibrozil, and CYP3A4 and CYP2C8 induction using rifampicin on the pharmacokinetics of SAR442168 in healthy male participants aged 18 to 45 years.

DETAILED DESCRIPTION:
Study duration per participant approximately 16 days for Cohort 1 and approximately 18 days for Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Male participant, between 18 and 45 years of age, inclusive.
* Body weight between 50.0 and 100.0 kg, inclusive, body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician. Participants with known hypersensitivity to any component of the IMP formulation or allergic disease diagnosed and treated by a physician.
* Any medication (including St John's Wort and ginseng) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Any contraindications to gemfibrozil or rifampicin, according to the applicable labelling.
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: AUClast of SAR442168 | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
  AUC up to the last measurable concentration
Pharmacokinetics: AUC of SAR442168 | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
  Area under the curve, reflects the concentration of drug

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration observed (Cmax) of SAR442168 | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
Pharmacokinetics: Cmax of SAR442168 metabolite(s) | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
Pharmacokinetics: AUC of SAR442168 metabolite(s) | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
Pharmacokinetics: Time to reach Cmax (tmax) of SAR442168 | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
Pharmacokinetics: tmax of SAR442168 metabolite(s) | Cohort 1: day1 period 1 to day 7 period 2; Cohort 2: day1 period 1 to day 9 period 2
Pharmacokinetics: Cmax of gemfibrozil | From Day 1 to Day 7 of Period 2
Pharmacokinetics: Cmax of gemfibrozil 1-O-glucuronide | From Day 1 to Day 7 of Period 2
Pharmacokinetics: tmax of gemfibrozil | From Day 1 to Day 7 of Period 2
Pharmacokinetics: tmax of gemfibrozil 1-O-glucuronide | From Day 1 to Day 7 of Period 2
Pharmacokinetics: Cmax of rifampicin | From Day 1 to Day 9 of Period 2
Pharmacokinetics: tmax of rifampicin | From Day 1 to Day 9 of Period 2
Numbers of participants with adverse events (AEs) | From baseline to End of Study (i.e. Period 2 Day 16 days in Cohort 1, and Period 2 Day18 days in Cohort 2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Prism Research-Site Number:8400001, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: INT16726 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25272&tenant=MT_SNY_9011